CLINICAL TRIAL: NCT06741540
Title: Effects of TDCS Intervention on Neoadjuvant Chemotherapy in Breast Cancer Patients with Mild to Moderate Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-1056
Record Dates: First submitted 2024-11-29; First posted 2024-12-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Neoadjuvant Chemotherapy; Depression; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Breast Neoplasms; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that modulates cortical excitability by applying a weak direct current through electrodes placed on the scalp. This technique usually lasts for 20-30 minutes and can affect brain function by altering cortical excitability, local cerebral blood flow, synaptic plasticity, and the balance of cortical excitation/inhibition. tDCS is widely used in clinical settings and has shown some clinical efficacy in treating common psychiatric and neurological disorders. It is also used to improve motor, perceptual, and cognitive processes, as well as to treat a variety of neurological and psychiatric diseases.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supportive psychotherapy group (No Intervention): Neoadjuvant chemotherapy with supportive psychotherapy and sham tDCS. A neoadjuvant chemotherapy regimen will be recommended to the patient based on the guidelines, combined with the patient's molecular typing and condition. Neoadjuvant chemotherapy lasts for 21 days per cycle, and the patient needs to be hospitalized for neoadjuvant chemotherapy once. During each neoadjuvant chemotherapy hospitalization, a full-time staff member will be arranged to perform sham tDCS treatment for the patient.
  The rest of the treatment was consistent with the tDCS group, but no current passed through the head-mounted device in this group.
  During the treatment，all patients in this group will recieve supportive psychotherapy, with mainly provide psychological support to patients.
- tDCS with supportive psychotherapy group (Experimental): Neoadjuvant chemotherapy with supportive psychotherapy and tDCS. A neoadjuvant chemotherapy regimen will be recommended to the patient based on the guidelines, combined with the patient's molecular typing and condition. Neoadjuvant chemotherapy lasts for 21 days per cycle, and the patient needs to be hospitalized for neoadjuvant chemotherapy once. During each neoadjuvant chemotherapy hospitalization, a full-time staff member will be arranged to perform tDCS treatment for the patient. The treatment is a head-mounted device, which is performed 1 hour before neoadjuvant chemotherapy and 2 hours after neoadjuvant chemotherapy. Each tDCS treatment lasts about 30 minutes. The patient's activities are not affected during the treatment, and no additional harm or pain is caused to the patient. A total of 6 tDCS treatments are completed per cycle of neoadjuvant chemotherapy, and 36 tDCS treatments will be completed during the entire treatment process.
  Interventions: Other: tDCS

INTERVENTIONS:
Other: tDCS — Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that modulates cortical excitability by applying a weak direct current through electrodes placed on the scalp. This technique usually lasts for 20-30 minutes and can affect brain function by altering cortical excitability, local cerebral blood flow, synaptic plasticity, and the balance of cortical excitation/inhibition.
  tDCS is widely used in clinical settings and has shown some clinical efficacy in treating common psychiatric and neurological disorders. It is also used to improve motor, perceptual, and cognitive processes, as well as to treat a variety of neurological and psychiatric diseases.
  Arms: tDCS with supportive psychotherapy group

SUMMARY:
Depression and anxiety are associated with higher incidence of tumors, cancer-specific mortality, and all-cause mortality.

Compared with patients with other types of cancer, breast cancer patients often accompany physical damage, changes in physiological status, decline in quality of life, sensitivity in interpersonal relationships, and side effects of drug treatment during the occurrence, development, and treatment of cancer, leading to long-term chronic mental stress. The prevalence of depression and anxiety in early-stage breast cancer patients in China is as high as 44.1% and 35.2%, respectively. A meta-analysis based on 282,203 breast cancer patients suggests that depression is related to breast cancer-specific mortality, and patients with breast cancer and depression have a poorer prognosis.

Intervention in response to stressors may improve psychological and physiological adaptation processes and even benefit quality of life and clinical health outcomes. More and more randomized controlled trials focus on improving the quality of life and adverse reactions of cancer patients after stress management, but there are few reports on the direct improvement of anti-tumor efficacy.

Therefore, we plan to conduct a small sample, exploratory, randomized controlled study to clarify the impact of transcranial direct current stimulation (tDCS) intervention on the efficacy of neoadjuvant chemotherapy in breast cancer patients with depressive symptoms. Newly diagnosed breast cancer patients will be assessed for emotions by mental health professionals, with a PHQ9 score of 5-14 and ≥ 5 symptoms considered positive, combined with enrollment criteria for screening. Patients who meet the enrollment criteria will be randomly divided into the control group (i.e., supportive psychotherapy group) and the experimental group (i.e., tDCS + supportive psychotherapy group). The primary study endpoint is the objective remission rate (ORR) of neoadjuvant treatment. This study aims to improve the depressive state of breast cancer patients undergoing neoadjuvant chemotherapy through physical therapy (tDCS) and to clarify whether there is a correlation between emotional intervention and neoadjuvant efficacy.

DETAILED DESCRIPTION:
Stress is the non-specific physiological and psychological response of the body to various stressors. Previous studies have proven that chronic stress is a recognized risk factor of tumors, participating in multiple stages such as tumor occurrence, development, metastasis, recurrence, and drug resistance. Epidemiological studies show that cancer patients often have chronic mental stress, accompanied by cognitive impairment, symptoms of depression and anxiety, and these patients have a poorer prognosis. Depression and anxiety are also associated with higher incidence of tumors, cancer-specific mortality, and all-cause mortality.

Breast cancer has become the most common malignant tumor in women, accounting for about 30% of new cancer cases in women. Since 1991, the mortality rate of breast cancer in women worldwide has slowed down due to the rapid development of screening and early diagnosis and treatment methods. It is worth noting that in China, breast cancer is still the leading cause of cancer in women, and its mortality rate is still on the rise. Compared with patients with other types of cancer, breast cancer patients often accompany physical damage, changes in physiological status, decline in quality of life, sensitivity in interpersonal relationships, and side effects of drug treatment during the occurrence, development, and treatment of cancer, leading to long-term chronic mental stress. The prevalence of depression and anxiety in early-stage breast cancer patients in China is as high as 44.1% and 35.2%, respectively. A meta-analysis based on 282,203 breast cancer patients suggests that depression is related to breast cancer-specific mortality, and patients with breast cancer and depression have a poorer prognosis.

Intervention in response to stressors may improve psychological and physiological adaptation processes and even benefit quality of life and clinical health outcomes. More and more randomized controlled trials focus on improving the quality of life and adverse reactions of cancer patients after stress management, but there are few reports on the direct improvement of anti-tumor efficacy.

This evidence proves that stress factors should not be ignored in the clinical process of tumor prevention and treatment. Our clinical practice has found that in addition to drug treatment, psychological and physical therapies are also effective for stress disorders. Therefore, we plan to conduct a small sample, exploratory, randomized controlled study to clarify the impact of transcranial direct current stimulation (tDCS) intervention on the efficacy of neoadjuvant chemotherapy in breast cancer patients with depressive symptoms. Newly diagnosed breast cancer patients will be assessed for emotions by mental health professionals, with a PHQ9 score of 5-14 and ≥ 5 symptoms considered positive, combined with enrollment criteria for screening. Patients who meet the enrollment criteria will be randomly divided into the control group (i.e., supportive psychotherapy group) and the experimental group (i.e., tDCS + supportive psychotherapy group). Both the experimental and control groups will receive supportive psychotherapy during the treatment process (mainly to provide psychological support for patients). The primary study endpoint is the objective remission rate (ORR) of neoadjuvant treatment, and the secondary study endpoints include pathological complete remission rate (pCR), improvement in depression scores (HAMD score changes), changes in breast-specific gamma imaging (BSGI), quality of life assessment after neoadjuvant chemotherapy, and ERP event-related potential detection. In addition, further exploratory research will be carried out, with stratified analysis based on breast cancer molecular typing, population characteristics, immune components, and changes in hormone levels.

This study aims to improve the depressive state of breast cancer patients undergoing neoadjuvant chemotherapy through physical therapy (tDCS) and to clarify whether there is a correlation between emotional intervention and neoadjuvant efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old;
* Newly diagnosed and pathologically confirmed breast cancer patients;
* Meet the guidelines for neoadjuvant chemotherapy indications, have no contraindications, and accept neoadjuvant treatment;
* At least one measurable lesion that can be assessed according to RECIST 1.1 criteria;
* Positive initial emotional assessment (5≤PHQ9 score ≤14), ≥ 5 symptoms and have not undergone other treatments;
* Cardiopulmonary function can withstand surgery, no other severe diseases, and Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
* Informed and willing to participate in the study, and have signed the informed consent form.

Exclusion Criteria:

* Concurrent severe physical illnesses;
* Suicidal tendencies;
* Pregnant or breastfeeding;
* Received tDCS physical therapy, systemic psychotherapy, antidepressant medication, or other treatments for negative emotions within the past 6 months;
* Patients with brain trauma and other organic brain diseases, and other contraindications for tDCS;
* Severe anxiety with GAD7 score ≥10.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | 18 weeks or 24 weeks, accroding to the neoadjuvant treatment completion
  Objective remission rate (ORR) of neoadjuvant treatment

SECONDARY OUTCOMES:
pathological complete remission rate (pCR) | 18 weeks or 24 weeks, after surgery completion, according to the neoadjuvant chemotherapy
  Pathological complete remission rate (pCR)
HAMD score changes | Evaluation was performed before and after neoadjuvant chemotherapy course (each course is 21 days)
  Improvement in depression scores (HAMD score changes)
BSGI | Every 2 cycles of neoadjuvant treatment (i.e., 6 weeks)
  Changes in breast-specific gamma imaging (BSGI)
QoL | 18 weeks or 24 weeks, accroding to the neoadjuvant treatment completion
  quality of life assessment after neoadjuvant chemotherapy, using the World Health Organization Quality of Life-brief Questionnaire (WHOQOL-BREF) .
ERP event-related potential detection | 18 weeks or 24 weeks, accroding to the neoadjuvant treatment completion
  Event-Related Potentials (ERP) are electrophysiological measures of the brain's electrical activity in response to specific events or stimuli, recorded via electroencephalography (EEG). They reflect cognitive processes and can be used to study various psychological phenomena with high temporal resolution, down to the millisecond. ERPs are valuable in clinical settings for assessing cognitive functions and are used in various fields, including psychiatry and neurology, to understand brain processing and diagnose conditions.

OTHER OUTCOMES:
Molecular typing of breast cancer | 18 weeks or 24 weeks, through neoadjuvant treatment completion
  Stratified analysis based on breast cancer molecular typing. Estrogen receptor (ER), progesterone receptor (PgR), Ki-67 labeling index and HER2 expression were evaluated by immunohistochemistry. A molecular subtype classification in five categories was adopted based upon the immunohistochemical assessment of ER, PgR, HER2 and Ki-67 according to the 2011 San Gallen consensus conference.
Population characteristics | 18 weeks or 24 weeks, through neoadjuvant treatment completion
  Information about population characteristics, including age, BMI, menstrual status, and previous medical conditions.
Immune components | Evaluation was performed at Day 1 of each course, up to 18 weeks or 24 weeks, through neoadjuvant treatment completion
  Tumor immune-related indicators in peripheral blood of patients, such as immune cell components, CRP, and cytokines (TNF-α, IL-6, IL-1, etc)
Hormone levels | Evaluation was performed at Day 1 of each course, up to 18 weeks or 24 weeks, through neoadjuvant treatment completion
  Stress-related hormones, such as thyroxine, cortisol, adrenocorticotropin, etc

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China